CLINICAL TRIAL: NCT06133153
Title: A Pivotal, Randomized, Subject- and Evaluator-blinded, Controlled, Non-inferiority, Multicenter, Parallel Group Comparison Study to Evaluate Effectiveness and Safety of THIODERM ELATE for Lip Augmentation in Order to Correct Lip Volume Deficit
Brief Title: THIODERM ELATE for Volume Augmentation in Lips
Acronym: TIVOLI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decision to change study design
Sponsor: Croma-Pharma GmbH (Industry)
Collaborators: Proinnovera GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPH-70602
Record Dates: First submitted 2023-11-03; First posted 2023-11-15 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Lip; Anomaly
Keywords: Lip Volume Deficit; Hyaluronic Acid Filler; Lip Augmentation; Dermal Filler
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Parallel-Group randomized study with a randomization ratio of 2:1 (Study Device : Comparator Device)
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinfolded during treatments; the blinded evaluating investigator will be blinded to device allocation and will have no access to unblinding information in the study files
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm THIODERM ELATE (Experimental): Subjects randomized to Arm A (approx. 66.7% of subjects) will receive THIODERM ELATE injected into both lips (Experimental Device) at the initial treatment and a potential touchup treatment.
  Interventions: Device: THIODERM ELATE
- Arm JUVÉDERM ULTRA (Active Comparator): Subjects randomized to Arm A (approx. 33.3% of subjects) will receive Juvéderm(R) Ultra injected into both lips (Comparator Device) at the initial treatment and a potential touchup treatment. .
  Interventions: Device: Juvéderm Ultra 3

INTERVENTIONS:
Device: THIODERM ELATE — Thiomer-crosslinked Hyaluronic Acid Dermal Filler with Lidocaine for Injection into Lips
  Arms: Arm THIODERM ELATE
Device: Juvéderm Ultra 3 — BDDE-crosslinked Hyaluronic Acid Dermal Filler with Lidocaine for Injection into Lips
  Arms: Arm JUVÉDERM ULTRA

SUMMARY:
A pivotal, randomized, subject- and evaluator-blinded, controlled, non-inferiority, multicenter, parallel group comparison study to evaluate effectiveness and safety of THIODERM ELATE for lip augmentation in order to correct lip volume deficit

DETAILED DESCRIPTION:
The clinical investigation will comprise randomization to one of two treatment groups:

* Test device: THIODERM ELATE
* Comparator device: Juvéderm® ULTRA 3 The Screening visit (Visit 1) will be performed within 2 weeks prior to randomization and will entail informed consent and screening assessments. During this visit the treating investigator will determine eligibility of subjects based on study inclusion and exclusion criteria - except for Baseline severity of lip volume deficit, that will be determined at Screening visit (Visit 1) by the blinded evaluator at the site using the 5-point LFS.

In addition, the subject's face will be photographed to document baseline condition for further assessments.

At Baseline visit (Visit 2 / Day 0), eligible subjects will be randomized in a 2:1 ratio and undergo lip augmentation treatment of both, upper and lower lip, with either THIODERM ELATE or Juvéderm® ULTRA 3 (baseline treatment).

If an optimal aesthetic correction has not been achieved after the baseline treatment as evaluated by the treating investigator, a touch-up treatment may be performed at Week 4 (Visit 3) using the same device as initially applied at Visit 2.

As of Week 36 (Visit 7 (SV1)) after last treatment (either baseline or touch-up treatment) of the initial treatment phase, subjects of both treatment groups (test device and comparator device) may qualify for a repeat-treatment, which will be done with THIODERM ELATE only. Further Screening visits for repeat-treatment may be conducted after Visit 7 (SV1) if the subject does not qualify at Visit 7(SV1) already for repeat-treatment.

Screening phase for repeat-treatment will be up to 20 weeks after Visit 7 (SV1) with Visit SV2 (12 weeks after Visit 7 (SV1)), Visit SV3 (16 weeks after Visit 7 (SV1)), and Visit SV4 (20 weeks after Visit 7 (SV1)).

As soon as the subject is eligible in LFS score as assessed by the blinded evaluator at the site, a full eligibility assessment for repeat-treatment will be done by the treating investigator. Subjects do not have to return to their baseline severity of lip volume deficit to be eligible and receive a repeat-treatment, but the present condition of lip volume deficit must meet the initial inclusion criterion (very thin lips or thin lips or moderately thick lips in both lips). The blinded evaluating investigator at the site decides if a subject is eligible for the repeat-treatment (regarding LFS).

Visit SV4 (20 weeks after Visit 7 (SV1)) will be the end of investigation visit for subjects who do not qualify for repeat-treatment. In case an inclusion criterion is not met / an exclusion criterion is met for repeat-treatment and further follow up in screening is not useful because the subject will apparently not qualify for repeat-treatment, the respective Screening Visit (SV1, SV2, SV3, or SV4) will be the end of investigation visit for the respective subject.

Subjects who are eligible and undergo repeat-treatment at Visit RT1 will enter the repeat-treatment follow-up phase. Subjects may receive a touch-up treatment after 4 weeks (Visit RT2) based on the treating investigator's judgement. The follow-up period will be 24 weeks after the last treatment (initial repeat treatment or touch-up treatment, respectively).

Follow-up visits on-site will occur at:

* Initial treatment phase: Week 4 and Week 8 after baseline treatment, and 12, 24, and 36 weeks after last treatment, i.e., baseline or touch-up treatment, respectively (Visits 3 to 7 (SV1))
* Screening phase for repeat-treatment: Week 12, 16 and 20 after Visit 7 (SV1) - (Visits SV2 to SV4)
* Repeat-treatment phase: Week 4, 8, 12, and 24 after initial repeat-treatment (Visits RT2 to RT5) regardless of whether a touch-up treatment has been performed or not (Visit RT2 to RT5) In addition to the on-site follow-up visits, 24-48 hours after each treatment the subjects will be contacted by phone for safety checkup. If applicable, the incidence, severity, seriousness, and type of adverse events resulting from device injection will be determined and closely followed up until resolution.

Lip volume deficit will be evaluated (live assessment) by the blinded evaluator at the site using the 5-point LFS during follow-up visits of the initial and repeat-treatment phase. In addition, volume change measurements will be done on 3D photographs.

Subject's pain perception during treatment and recovery from treatment will be evaluated by means of a numerical pain rating scale (NPRS) immediately after, and 15 and 30 minutes after last injection of each treatment session.

Global aesthetic improvement will be evaluated by reviewing and comparing current photographs relative to photographs taken at Screening visit. Both - the blinded evaluator at the site and the subject - will assess the global aesthetic improvement (using the modified GAIS) at each on-site visit after subject was fully treated (baseline and touch-up treatment, as applicable) during the initial treatment phase.

Subject´s satisfaction with the outcome of the treatment will be assessed with the FACE-QTM questionnaires "Satisfaction with Outcome" and "Satisfaction with Lips" at each on-site visit after subject was fully treated (baseline / repeat-treatment and touch-up treatment, as applicable) during the initial and repeat-treatment phase, respectively. Subject´s "Satisfaction with Lips" will also be assessed at Visit 2 (Baseline visit) and Visit RT1.

The safety will be evaluated based on occurrence of adverse events, which will be collected at each visit (on-site and telephone visits) throughout the clinical investigation, beginning after signature of the ICF until the last visit.

To identify potential adverse events post-administration a safety evaluation after 30 minutes needs to take place.

A subject diary will be used to record injection site reactions, and symptoms of interest (i.e., vaso-occlusive events, such as changes in vision or symptoms of stroke) over the first four weeks (28 days) after each treatment (i.e., either 4 weeks after baseline and repeat-treatment or in total 8 weeks in case of touch-up treatment).

To evaluate any potential vision changes, visual examinations (including Snellen visual acuity, confrontational visual fields and ocular motility) will be additionally performed at treatment visits (prior to- and 30 min after any treatment) and at all follow-up visits of the initial and repeat-treatment phase. A basic neurological examination (F.A.S.T) will be performed for all subjects who show signs of ophthalmic complications due to filler injection.

Abnormal clinically significant changes in visual examination or experience of neurological symptoms indicative of a vaso-occlusive event after any treatment will lead to withdrawal of the subject from further treatment(s) in case an eye specialist or neurologist confirms that the result is related to a vascular injection of the dermal filler. The subjects may remain in the study for at least safety assessments during the scheduled study visits. In such case, stopping the entire investigation will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects aged 18-75 years (inclusive) of age at Screening (Visit 1).

2. Subjects with approximately symmetric moderate to severe lip volume deficit (severity scores of 1, 2, or 3 on the 5-point Lip Fullness Scale), as assessed by the blinded evaluator at the site. Approximately symmetric is defined as a maximum of 1 grade difference between upper and lower lip. Both lips need to meet the eligibility criterion of severity score 1, 2 or 3 on the 5-point LFS.

3. Females of childbearing potential must have a negative urine pregnancy test and must agree to use a highly effective method of birth control throughout the entire investigation.

Male subjects with female partners of child-bearing potential must agree to use contraception throughout the entire study (surgical sterilization or a physical barrier such as a condom).

4. Healthy skin in and around the treatment area and free of diseases that could interfere in the effectiveness assessments.

5. Intact or permanently replaced incisor and canine teeth in the upper and lower jaw.

6. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of the entire investigation.

7. Subjects who understand the purpose and conduct of the study and having given written informed consent and are willing and able to attend the study visits as judged by the treating investigator.

Exclusion Criteria:

Subjects who meet ANY of the following criteria are NOT eligible for the clinical investigation and must not be enrolled:

1. Females, who are pregnant and/or, lactating or planning to become pregnant during the clinical investigation.
2. History of allergy or hypersensitivity to hyaluronic acid preparations, lidocaine or any amide-based anesthetic.
3. Prior surgery, scars or tattoo to the upper or lower lip or lip line; surgery and tattooing are prohibited until end of clinical investigation.
4. Tooth gap, overbite, beard longer three-day beard, or excessive facial hair that could interfere in evaluation of treatment as judged by the treating investigator.

   Note: If subject agrees to shave beard, incl. three-day beard, or excessive facial hair prior to on-site visits, the subject is eligible for the investigation.
5. Presence of any abnormal lip structure, such as a scar or lump or severe lip asymmetry, as judged by the treating investigator.
6. Presence of infectious, inflammatory or proliferative cancerous or pre-cancerous lesions in the treatment area.
7. Re-current (at least three times over the last year) herpes simplex in the treatment area.
8. History or presence of the following autoimmune or connective tissue diseases: Scleroderma, advanced Lupus erythematosus that is unstable, acute rheumatic fever with heart complications.
9. AIDS that is not well controlled as determined by the treating investigator.
10. Uncontrolled (or unstable) Diabetes mellitus or uncontrolled / unstable other systemic diseases as per treating investigator discretion.
11. Implantation of HA or collagen dermal fillers in the treatment area within the preceding 18 months prior to Screening (Visit 1) and during the entire investigation.
12. Previous permanent implant or treatment with non-HA or non-collagen filler in or around the lip area (including lips, oral commissures, nasolabial folds, marionette, and perioral lines) and until end of the investigation.
13. Previous botulinum toxin treatment in or around the lip area (including lips, oral commissures, nasolabial folds, marionette, and perioral lines) within 12 months before Screening (Visit 1) and until end of clinical investigation.
14. Previous facial plastic surgery, tissue augmentation with silicone, fat or another non-absorbable substance (permanent fillers) and semi-permanent / long-lasting fillers (e.g., poly-L-lactic acid (PLLA), Polymethylmethacrylate (PMMA) filler) or non-absorbable sutures in the area of device application and during the entire investigation.
15. Subject has received any of the following treatments:

    * Full ablative facial laser therapy,
    * Absorbable sutures (threads) in the treatment area,
    * Facial lipolysis, including submental fat treatments or
    * Bariatric surgery within the last 12 months prior to Screening (Visit 1) or is planning to undergo such procedures during entire investigation.
16. Subject has received dermabrasion, mesotherapy, chemical peeling, or micro-needling in the face within 30 days prior to baseline treatment and touch-up treatment.
17. The use of the following anticoagulant or thrombolytic medications is not allowed from ten days pre- to three days post injection (baseline treatment):

    * Vitamin K Antagonists (e.g., Warfarin)
    * Oral Direct Factor Xa Inhibitors (e.g., Apixaban, Betrixaban, Edoxaban, Rivaroxaban)
    * Oral Direct Factor IIa Inhibitors (e.g., Dabigatran)
18. Planned dental/oral surgery or modification (bridge-work, implants) within four weeks prior to each injection and to a minimum of four weeks post injection baseline treatment and touch-up treatment.
19. Subjects who have one of the following assessments during the visual examinations at Screening (Visit 1): Snellen visual acuity test worse than 20/40 (with corrective eyewear, if applicable), abnormal confrontational visual field test, or abnormal ocular motility test.
20. Any medical condition prohibiting the inclusion in the study according to the judgment of the treating investigator.
21. Previous enrollment in this clinical investigation.
22. Current participation in another clinical trial, or treatment with any investigational drug/medical device within 30 days prior to Screening (Visit 1) or within five half-lives of an investigational drug, whichever is longer and during the entire investigation.
23. Subjects who experienced fat loss for a minimum of 10% of body weight over the last 12 months (e.g., post bariatric patients), or subjects who have the intention to change eating habits that result in a weight gain or loss ≥10% during the entire investigation.
24. Any individual whose willingness to volunteer in this clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants).
25. Close affiliation with the investigator (e.g., a close relative, financially dependent on the study site) or subject who is an employee of the sponsor's company or group companies of the Sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Lip Volume from Baseline | Week 12
  Changes from baseline in LFS scores of the upper and lower lips based on the blinded evaluator´s live assessment at Week 12 after last injection of initial treatment phase.

SECONDARY OUTCOMES:
Subject's assessment of Aesthetic Improvement | Week 12
  Improvement over baseline ("much improved" or "improved"), based on the subject's assessment at Week 12 after last injection of initial treatment phase using the 5-point modified GAIS.
Response Rate | Weeks 8, 24, and 36.
  Responder status, based on the blinded evaluator´s live assessment on the 5-point LFS at Week 8, 24, and 36 after last injection of initial treatment phase compared to the score at Baseline visit.
Change in Lip Volume from Baseline | Weeks 8, 24, and 36.
  Change of lip volume deficit measured on the 5-point LFS and based on the blinded evaluator´s live assessment at Week 8, 24, and 36 after last injection of initial treatment phase compared to the score at Baseline visit.
Global Aesthetic Improvement over baseline - Subject | Weeks 8, 24, and 36.
  Improvement over baseline ("much improved" or "improved"), based on subject´s assessment at Week 8 after baseline and weeks 24 and 36 after last injection of initial treatment phase using the 5-point modified GAIS.
Global Aesthetic Improvement over baseline - Blinded Evaluator | Weeks 8, 24, and 36.
  Improvement over baseline ("much improved" or "improved"), based on the blinded evaluator's assessment at Week 8 after baseline and weeks 12, 24, and 36 after last injection of initial treatment phase using the 5-point modified GAIS.
Subject Satisfaction - Face-Q(TM) Outcome | Weeks 8, 12, 24, and 36.
  The extent of subject´s satisfaction with overall treatment outcome at Week 8 after baseline and weeks 12, 24, and 36 after last injection of initial treatment phase as assessed by the subject using the Face-QTM Questionnaire "Satisfaction with Outcome".
Subject Appearance Appraisal - Face-Q(TM) Satisfaction with Lips | Weeks 8, 12, 24, and 36.
  The extent of subject´s appearance appraisal at Week 8 after baseline and weeks 12, 24, and 36 after last injection of initial treatment phase as assessed by the FACE-QTM questionnaire "Satisfaction with Lips" compared to Baseline visit.
Pain Assessment | Day 0; Week 4
  Subject evaluation of pain after each treatment (repeat and touch-up-treatment) on an 11-point numerical pain rating scale (NPRS), where 0 is no pain and 10 is the worst pain imaginable
Injection Volume | Day 0; Week 4
  Injection volume required to achieve optimal aesthetic result at each treatment (initial and touch-up treatment together)

OTHER OUTCOMES:
Safety Endpoint: Adverse Events | through study completion, an average of 36 Weeks
  Adverse events during the entire study period including repeat-treatment phase (long-term safety). Other symptoms of interest will be recorded in subject diary during the first 4 weeks (28 days) after each treatment (i.e., either 4 weeks after baseline and repeat-treatment and in total 8 weeks in case of touch-up treatment) and documented as AE by investigator.
Safety Endpoint: Injection Site Reactions (ISR) | Day 0; Week 4
  4 weeks (28 days) after each treatment (i.e., either 4 weeks after baseline and repeat-treatment and in total 8 weeks in case of touch-up treatment). Injection site reactions will be assessed overall and for each lip (i.e., upper and lower lips separately).

CONTACTS AND LOCATIONS:
Locations (1):
- H&P Ambulatorien GmbH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No